CLINICAL TRIAL: NCT06254144
Title: Neuroimaging Study for Decoding Emotional States and Identifying Neural Circuits to Disengage From Negative Thinking
Acronym: RNT-decoding
Status: Enrolling by invitation | Type: Observational
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-006
Record Dates: First submitted 2024-01-26; First posted 2024-02-12 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: functional magnetic resonance imaging (fMRI) — The investigators will utilize standard BOLD fMRI in blocked-design tasks and resting state (participant is given no overt task) in the study. Anatomical scans with T1-weighted contrast, quantitative measurement of spin relaxation times, and diffusion tensor imaging (DTI) are also used as an anatomical reference for functional activation as well as to investigate a brain structural relationship with the participants' task performance, including successful emotion regulation.

SUMMARY:
The purpose of this study is to decode different thinking states from the brain activation patterns and identify the neural circuits that disengage from these thinking patterns using functional magnetic resonance imaging (fMRI) measurement in individuals with major depressive disorder.

DETAILED DESCRIPTION:
This study aims to identify brain activation patterns associated with successful disengagement from negative thinking for MDD-affected participants. The investigators will use a machine learning classifier to decode thinking states from participants' fMRI signals. The decoder is utilized to trace the thinking state's time course as a measure of regulation performance. Investigating the brain activation correlated with the time course of the regulation success can indicate the neural circuits contributing to disengaging from negative thinking. The investigators will also explore the most effective regulation strategy for individual participants. Participants will be instructed to use three regulation strategies: mindfulness by focusing on breathing, distraction with positive thinking, and reinterpretation of a negative thing in a positive way. The investigators expect that the effective strategy could vary across participants, which could be associated with the variability of brain activation patterns in negative thinking.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and complying with protocol requirements.
* Participants who are fluent and literate in English and are able to understand and provide written, informed consent and any required privacy authorization prior to the initiation of any study procedures.
* Male or female, 18 to 65 years.
* Current diagnosis of MDD who are currently depressed defined by the MINI.
* Participants who have moderate depressive symptoms (Patient Health Questionnaire: PHQ-9 ≥ 10 or Quick Inventory of Depressive Symptomatology: QIDS-SR ≥ 11).

Exclusion Criteria:

* Diagnosis of Schizophrenia spectrum or other psychotic disorders.
* Bipolar I Disorder.
* Active suicidal ideation with a plan and intent or suicidal ideation/attempts in the past 6-12 months.
* Current diagnosis of post-traumatic disorder (PTSD) defined by the MINI.
* Change in the dose or prescription of medication within the 6 weeks before enrolling in the study that could affect brain functioning.
* Moderate to severe substance use disorder within the last 12 months.
* A positive test for drugs of abuse, including but not limited to alcohol (breath test), cocaine, marijuana, opiates, amphetamines.
* Use of > 400 mg caffeine or nicotine within the past 2 hours. Medical Conditions
* History of unstable liver or renal insufficiency.
* Significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, hematologic, rheumatologic, or metabolic disturbance.
* Moderate to severe traumatic brain injury or neurocognitive disorders with evidence of neurological deficits.
* Co-morbid medical conditions, including cardiovascular (e.g., history of acute coronary events, stroke) and neurological diseases (e.g., Parkinson's, epilepsy).
* Co-morbid inflammatory disorders (e.g., rheumatoid arthritis, autoimmune disorders).
* Uncontrolled or unstable medical conditions deemed risky by investigators.
* Chronic or acute infectious illness (e.g., HIV, SARS-CoV-2).
* Current use of hormone-containing medications (excluding contraceptives), immunosuppressive medications, non-steroid anti-inflammatory drugs, or analgesics.

MRI Contraindications

* Contraindications for MRI (e.g., metal fragments, cardiac pacemaker). Miscellaneous
* Unwillingness or inability to complete any of the major aspects of the study protocol.
* Non-correctable vision or hearing problems.
* Lack of understanding of English.
* BMI > 40 or < 18.5.
* Pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with major depressive disorders
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Classification accuracy of different internal thoughts | 2 weeks
  fMRI brain images captured during various internal thought processes are used as input to a machine learning classifier. This classifier is trained to discriminate between different mental states. In this context, "classification accuracy" refers to the classifier's ability to accurately identify or predict the specific mental state based on the fMRI data. This measures the classifier's effectiveness in differentiating between mental states by analyzing patterns of brain activity. Classification accuracy is assessed using the area under the receiver operating characteristic curve (AUC), which is robust to imbalances in sample size for each mental state by incorporating the relationship between true positive and false positive rates. A higher AUC indicates better classifier performance.
Changes in blood oxygen level-dependent (BOLD) signals across the whole brain during different internal thoughts and emotion regulation strategies. | 2 weeks
  Differences in whole brain activation patterns, elicited by various internal thoughts and emotion regulation strategies, will be quantified based on changes in blood oxygen level-dependent (BOLD) signals in the whole brain. An increase in BOLD signal indicates a greater brain activation.

OTHER OUTCOMES:
Correlations of Ruminative Responses Scale (RRS) Brooding subscores with classification accuracy and BOLD signal changes | 2 weeks
  The RRS Brooding subscale is a self-report scale to measure brooding ruminative responses. A higher score indicates higher brooding ruminative responses with a maximum score of 20 and a minimum score of 5.
  Classification accuracy and whole brain activation pattern differences in BOLD signals from brain imaging will be correlated with the RRS Brooding subscale.
Correlations of Ruminative Responses Scale (RRS) Depression subscores with classification accuracy and BOLD signal changes | 2 weeks
  The RRS Depression subscale is a self-report scale to measure depressive ruminative responses. A higher score indicates higher ruminative responses with a maximum score of 48 and a minimum score of 12.
  Classification accuracy and whole brain activation pattern differences in BOLD signals from brain imaging will be correlated with the RRS Depression subscale.
Correlations of Ruminative Responses Scale (RRS) Reflection subscores with classification accuracy and BOLD signal changes | 2 weeks
  The RRS Reflection subscale is a self-report scale to measure reflective ruminative responses. A higher score indicates higher ruminative responses with a maximum score of 20 and a minimum score of 5.
  Classification accuracy and whole brain activation pattern differences in BOLD signals from brain imaging will be correlated with the RRS Reflection subscale.
Correlations of Ruminative Responses Scale (RRS) total score with classification accuracy and BOLD signal changes | 2 weeks
  The RRS is a self-report scale to measure ruminative responses. A higher score indicates higher ruminative responses with a maximum score of 88 and a minimum score of 22.
  Classification accuracy and whole brain activation pattern differences in BOLD signals from brain imaging will be correlated with the RRS total scores.
Correlations of Montgomery-Asberg Depression Rating Scale (MADRS) scores with classification accuracy and BOLD signal changes | 2 weeks
  The MADRS is an interviewer-rated scale to measure the severity of depressive symptoms. A higher score indicates severer depression with a maximum score of 60 and a minimum score of 0.
  Classification accuracy and whole brain activation pattern differences in BOLD signals from brain imaging will be correlated with the MADRS scores.
Correlations of Hamilton Anxiety Rating Scale (HAM-A) scores with classification accuracy and BOLD signal changes | 2 weeks
  The HAMA is an interviewer-rated scale to measure the severity of anxiety symptoms. A higher score indicates severer anxiety with a maximum score of 56 and a minimum score of 0.
  Classification accuracy and whole brain activation pattern differences in BOLD signals from brain imaging will be correlated with the HAM-A scores.
Correlations of Brief State Rumination Inventory (BSRI) scores with classification accuracy and BOLD signal changes | 2 weeks
  The BSRI is a self-report scale to measure state rumination. A higher score indicates higher state rumination with a maximum score of 800 and the minimum score of 0.
  Classification accuracy and whole brain activation pattern differences in BOLD signals from brain imaging will be correlated with the BSRI scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No